CLINICAL TRIAL: NCT03408392
Title: An Open-label, Randomised, Single-dose, Two-period Cross-over Study to Evaluate Bioequivalence of SKF101804 Cefixime 200 mg/5 mL Suspension Versus Cefixime 200 mg/5 mL Suspension Reference Product in Healthy Adult Participants Under Fasting Conditions
Brief Title: Bioequivalence Study Between SKF101804 Cefixime 200 Milligram (mg)/5 Milliliter (mL) Suspension Versus Cefixime 200 mg/5 mL Suspension Reference Product in Healthy Adult Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205731
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Results first posted 2019-03-22 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Infections, Bacterial
Keywords: Single dose; Oral suspension; Bioequivalence; Cefixime; Two-way crossover
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test followed by Reference Formulation (Experimental): Subjects will be randomized to receive single dose of Test formulation (SKF101804: cefixime 200 mg/ 5 mL) on Day 1 of the treatment period 1 and Reference formulation (cefixime 200 mg/5 mL) on Day 1 of the treatment period 2. There will be wash out period of 7-14 days between the two treatment periods.
  Interventions: Drug: Test formulation A; Drug: Reference formulation B
- Reference followed by Test Formulation (Experimental): Subjects will be randomized to receive single dose of Reference formulation (cefixime 200 mg/5 mL) on Day 1 of the treatment period 1 and Test formulation (SKF101804: cefixime 200 mg/ 5 mL) on Day 1 of the treatment period 2. There will be wash out period of 7-14 days between the two treatment periods.
  Interventions: Drug: Test formulation A; Drug: Reference formulation B

INTERVENTIONS:
Drug: Test formulation A — Test formulation: SKF101804 will be available as oral suspension supplied as powder for reconstitution (Off-white to cream coloured powder). Subjects will receive single dose of 5 mL of suspension thus receiving 200 mg dose of cefixime. The suspension is a white to off white viscous suspension with a fruit flavor and odor.
Drug: Reference formulation B — Reference formulation will be available as oral suspension supplied as powder for reconstitution (Off-white to cream coloured powder). Subjects will receive single dose of 5 mL of suspension thus receiving 200 mg dose of cefixime. The suspension is a white to off white viscous suspension with a strawberry flavor and odor.

SUMMARY:
This study is open-label, randomized two-way cross-over study to determine if cefixime 200 mg/5 mL powder for suspension (test formulation: SKF101804) is bioequivalent to cefixime 200 mg/5 mL suspension reference formulation. Study will be conducted in 28 healthy adult subjects under fasting conditions. There will be two treatment periods and each subject will participate in both periods. The washout period between both treatment periods will be 7-14 days. Subjects will be randomized to either of treatment sequences of reference followed by test or test followed by reference to receive a single dose of test or reference formulation on Day 1 in each treatment period. The study will last for 5 to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Subject must be healthy, non-smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included at investigator discretion in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subject with a body weight 50 kilogram (kg) and body mass index (BMI) within the range 19-30 kilogram per meter square (kg/m^2) (inclusive).
* A healthy male subject must agree to use contraception during the treatment period and for at least 5 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.
* A subject should be capable of giving signed informed consent.

Exclusion Criteria:

* Subject with history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Subjects with any other condition that is capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Subject with abnormal renal function, as determined by creatinine clearance and considered as clinically significant by the investigator will be excluded.
* Subject with abnormal blood pressure (BP) as determined by the investigator.
* Subject with lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Subject who had breast cancer within the past 10 years.
* ALT >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Subject with current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subject with history of colitis
* Subject with history of cephalosporin induced hemolytic anemia.
* QT interval corrected for heart rate according to Bazett's formula (QTcB) >450 milliseconds (msec). Subjects with a known risk of QT prolongation will be excluded.
* Past or intended use of over-the-counter or prescription medication including herbal medications, within 14 days prior to dosing unless in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 90 days.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 90 days before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Presence of Hepatitis B surface antigen (HBsAg) at screening. Positive Hepatitis C antibody test result at screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) test is obtained.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Subjects with regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Subjects with urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Subjects who are sensitive to heparin or heparin-induced thrombocytopenia.
* Subjects with known sensitivity to any drugs from the class of cephalosporin, or components thereof.
* Subjects with known sensitivity to any drugs from the class of penicillin, or components thereof.
* Subjects with known sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, single-dose, two-period cross-over study to evaluate bioequivalence of SKF101804 Cefixime 200 milligram (mg)/5 milliliter (mL) suspension versus Cefixime 200 mg/5 mL suspension reference product in healthy adult participants under fasting conditions. Participants were enrolled at a single center in South Africa.
Pre-assignment Details: Participants received treatment in one of the two sequences; SKF101804 cefixime 200mg/5mL suspension (Test formulation) followed by cefixime 200mg/5mL suspension (Reference formulation)or vice versa in each of the treatment period 1 and 2. A total number of 28 participants were randomized.
Groups:
- SKF101804 Cefixime Followed by Cefixime Reference Formulation: Eligible participants received single dose of Test formulation (SKF101804 cefixime 200 mg /5 mL suspension) orally on Day 1 in Treatment period 1. It was followed by a washout period of at least 7 days and not more than 14 days. Participants received single dose of Reference formulation (cefixime 200 mg/5 mL suspension) orally on Day 1 in Treatment period 2.
- Cefixime Reference Formulation Followed by SKF101804 Cefixime: Eligible participants received single dose of Reference formulation (cefixime 200 mg/5 mL suspension) orally on Day 1 in Treatment period 1. It was followed by a washout period of at least 7 days and not more than 14 days. Participants received single dose of Test formulation (SKF101804 cefixime 200 mg /5 mL suspension) orally on Day 1 in Treatment period 2.
Period: Treatment Period 1 (16 Days)
Arm/Group | SKF101804 Cefixime Followed by Cefixime Reference Formulation | Cefixime Reference Formulation Followed by SKF101804 Cefixime
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Wash-out Period (14 Days)
Arm/Group | SKF101804 Cefixime Followed by Cefixime Reference Formulation | Cefixime Reference Formulation Followed by SKF101804 Cefixime
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Treatment Period 2 (16 Days)
Arm/Group | SKF101804 Cefixime Followed by Cefixime Reference Formulation | Cefixime Reference Formulation Followed by SKF101804 Cefixime
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Eligible participants received a single dose of Test formulation (SKF101804 cefixime 200 mg /5 mL suspension) followed by Reference formulation (cefixime 200 mg/5 mL suspension) or vice versa, administered orally on Day 1 in each treatment period 1 and 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mixed Race | 3
  White/Caucasian/European Heritage | 4
  Black or African American | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments (AUC [0-t]) for Cefixime
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of cefixime under fasted state. Pharmacokinetic analysis of cefixime was conducted using non-compartmental methods. Pharmacokinetic Population comprised of participants who completed the study and for whom primary pharmacokinetic parameters could be calculated for all treatment periods were included in the statistical pharmacokinetic analysis of the study.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0 8.0, 10.0, 12.0, 16.0 and 20.0 hours post dose on Day 1, 24.00 hours post dose on Day 2 of each treatment period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Groups:
- SKF101804 Cefixime: Eligible participants received SKF101804 cefixime 200mg/5mL suspension (Test formulation), administered orally on Day 1 in each treatment period 1 or 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
- Cefixime Reference Formulation: Eligible participants received Cefixime 200mg/5mL suspension (Reference formulation), administered orally on Day 1 in each treatment period 1 or 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Hour*nanogram per milliliter | 20000 (32.9) | 19000 (34.3)
Statistical Analysis 1: Comparison: SKF101804 Cefixime vs Cefixime Reference Formulation; Test type: Equivalence — Bio-equivalence analysis comparing cefixime test and reference product has been presented; Percentage ratio = 105.38, 90% CI 2-sided [96.11 to 115.54]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Within a Participant Across All Treatments of Cefixime
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of cefixime under fasted state. Pharmacokinetic analysis of cefixime was conducted using non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Nanogram per milliliter | 2670 (29.4) | 2640 (30.5)
Statistical Analysis 1: Comparison: SKF101804 Cefixime vs Cefixime Reference Formulation; Test type: Equivalence — Bio-equivalence analysis comparing cefixime test and reference product has been presented; Percentage ratio = 101.14, 90% CI 2-sided [93.37 to 109.55]

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to (AUC [0-infinity]) Across All Treatments for Cefixime
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Hour*nanogram per milliliter | 20700 (31.8) | 19700 (33.3)
Statistical Analysis 1: Comparison: SKF101804 Cefixime vs Cefixime Reference Formulation; Test type: Equivalence — Bio-equivalence analysis comparing cefixime test and reference product has been presented; Percentage ratio = 105.14, 90% CI 2-sided [96.31 to 114.78]

4. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for Cefixime
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of cefixime under fasted state. Pharmacokinetic analysis of ciprofloxacin was conducted using non-compartmental methods. Tmax of cefixime was analyzed using a nonparametric test to compute point estimate of the median and full range.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Hours | 4.005 [2.50 to 6.02] | 4.005 [2.02 to 4.51]

5. Secondary Outcome: Percentage of AUC(0-infinity) Obtained by Extrapolation (%AUCex) for Cefixime
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Percentage of AUCex | 3.24 (51.4) | 3.32 (67.8)

6. Secondary Outcome: Terminal Phase Half-life (T1/2) for Cefixime
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Hours | 3.18 (15.0) | 3.13 (14.7)

7. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect or other situations. The analysis was performed on Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment. Participants were analyzed according to the treatment they actually received.
Time Frame: Up to Day 16 in each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 28 | 28
Participants
  Non-serious AEs | 0 | 0
  SAEs | 0 | 0

8. Secondary Outcome: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), and Aspartate Aminotransferase (AST) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including ALT, ALP and AST.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Units per liter
  ALT; Period 1; Day -1, 24 Hours Pre-dose | 16.6 (10.23) | 15.6 (5.67)
  ALT; Period 1; Day 2, 24 Hours Post-dose | 13.6 (7.09) | 14.0 (5.76)
  ALT; Period 2; Day -1, 24 Hours Pre-dose | 16.4 (8.98) | 16.7 (9.15)
  ALT; Period 2; Day 2, 24 Hours Post-dose | 14.1 (7.07) | 14.9 (7.68)
  ALP; Period 1; Day -1, 24 Hours Pre-dose | 80.4 (12.85) | 74.8 (18.25)
  ALP; Period 1; Day 2, 24 Hours Post-dose | 75.5 (14.27) | 67.1 (15.23)
  ALP; Period 2; Day -1, 24 Hours Pre-dose | 72.4 (17.58) | 80.9 (15.81)
  ALP; Period 2; Day 2, 24 Hours Post-dose | 69.7 (16.96) | 76.9 (15.13)
  AST; Period 1; Day -1, 24 Hours Pre-dose | 20.9 (4.40) | 20.6 (4.22)
  AST; Period 1; Day 2, 24 Hours Post-dose | 16.7 (2.64) | 17.1 (3.45)
  AST; Period 2; Day -1, 24 Hours Pre-dose | 20.5 (6.00) | 19.9 (4.57)
  AST; Period 2; Day 2, 24 Hours Post-dose | 16.8 (3.75) | 17.8 (4.08)

9. Secondary Outcome: Blood Urea Nitrogen (BUN) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of BUN.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Milligrams per deciliter
  Period 1; Day -1, 24 Hours Pre-dose | 10.354 (1.972) | 10.300 (4.120)
  Period 1; Day 2, 24 Hours Post-dose | 12.945 (2.349) | 12.258 (2.664)
  Period 2; Day -1, 24 Hours Pre-dose | 10.841 (3.571) | 11.844 (2.017)
  Period 2; Day 2, 24 Hours Post-dose | 12.041 (2.166) | 12.796 (1.599)

10. Secondary Outcome: Calcium, Glucose, Potassium and Sodium at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including calcium, glucose, potassium and sodium.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Millimoles per liter
  Calcium;Period 1;Day -1, 24 Hours Pre-dose | 2.393 (0.059) | 2.399 (0.134)
  Calcium;Period 1;Day 2, 24 Hours Post-dose | 2.308 (0.068) | 2.304 (0.076)
  Calcium;Period 2;Day -1, 24 Hours Pre-dose | 2.364 (0.099) | 2.376 (0.060)
  Calcium;Period 2;Day 2, 24 Hours Post-dose | 2.351 (0.087) | 2.378 (0.081)
  Glucose;Period 1;Day -1, 24 Hours Pre-dose | 4.684 (0.256) | 4.616 (0.267)
  Glucose;Period 1;Day 2, 24 Hours Post-dose | 4.728 (0.229) | 4.676 (0.295)
  Glucose;Period 2;Day -1, 24 Hours Pre-dose | 4.521 (0.347) | 4.571 (0.404)
  Glucose;Period 2;Day 2, 24 Hours Post-dose | 4.851 (0.375) | 4.812 (0.278)
  Sodium;Period 1;Day -1, 24 Hours Pre-dose | 143.86 (1.460) | 145.00 (1.414)
  Sodium;Period 1;Day 2, 24 Hours Post-dose | 141.07 (1.439) | 141.43 (1.604)
  Sodium;Period 2;Day -1, 24 Hours Pre-dose | 141.21 (1.251) | 141.50 (1.912)
  Sodium;Period 2;Day 2, 24 Hours Post-dose | 139.43 (1.089) | 139.64 (1.550)
  Potassium;Period1;Day -1, 24 Hours Pre-dose | 4.634 (0.457) | 4.404 (0.316)
  Potassium;Period1;Day 2, 24 Hours Post-dose | 4.522 (0.444) | 4.286 (0.206)
  Potassium;Period 2;Day -1, 24 Hours Pre-dose | 4.371 (0.220) | 4.521 (0.346)
  Potassium;Period 2;Day 2, 24 Hours Post-dose | 4.269 (0.334) | 4.555 (0.402)

11. Secondary Outcome: Total Bilirubin (Total Bil), Direct Bilirubin (Direct Bil) and Creatinine (Creat) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including total bil, direct bil and creat.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Micromoles per liter
  Creat; Period 1; Day -1, 24 Hours Pre-dose | 82.4 (15.29) | 83.4 (15.45)
  Creat; Period 1; Day 2, 24 Hours Post-dose | 79.9 (12.00) | 85.9 (15.59)
  Creat; Period 2; Day -1, 24 Hours Pre-dose | 81.1 (14.31) | 78.5 (14.21)
  Creat; Period 2; Day 2, 24 Hours Post-dose | 83.9 (15.33) | 78.4 (12.71)
  Total bil; Period1;Day -1, 24 Hours Pre-dose | 10.14 (4.633) | 10.99 (6.235)
  Total bil; Period1;Day 2, 24 Hours Post-dose | 6.83 (3.004) | 8.10 (6.191)
  Total bil; Period2;Day -1, 24 Hours Pre-dose | 9.90 (7.205) | 8.22 (3.516)
  Total bil; Period2;Day 2, 24 Hours Post-dose | 6.47 (3.749) | 6.16 (2.843)
  Direct bil; Period1;Day -1, 24 Hours Pre-dose | 3.68 (1.294) | 4.01 (1.794)
  Direct bil; Period1;Day 2, 24 Hours Post-dose | 2.65 (0.959) | 2.93 (1.630)
  Direct bil; Period2;Day -1, 24 Hours Pre-dose | 3.58 (1.945) | 3.12 (1.057)
  Direct bil; Period2;Day 2, 24 Hours Post-dose | 2.55 (1.149) | 2.49 (0.972)

12. Secondary Outcome: Total Protein at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of total Protein.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Grams per liter
  Period 1; Day -1, 24 Hours Pre-dose | 74.34 (3.354) | 74.77 (4.725)
  Period 1; Day 2, 24 Hours Post-dose | 67.90 (3.295) | 67.97 (2.635)
  Period 2; Day -1, 24 Hours Pre-dose | 73.76 (3.995) | 72.57 (3.886)
  Period 2; Day 2, 24 Hours Post-dose | 67.64 (3.181) | 67.89 (4.211)

13. Secondary Outcome: Platelets, Neutrophils, Monocytes, Lymphocytes, Leucocyte, Eosinophils and Basophils at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematology parameters including platelets, neutrophils, monocytes, lymphocytes, leucocyte, eosinophils and basophils.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
10^9 cells per liter
  Basophil; Period 1;Day -1, 24 Hours Pre-dose | 0.023 (0.017) | 0.022 (0.013)
  Basophil; Period 1;Day 2, 24 Hours Post-dose | 0.024 (0.012) | 0.025 (0.011)
  Basophil; Period 2;Day -1, 24 Hours Pre-dose | 0.026 (0.012) | 0.029 (0.025)
  Basophil; Period 2;Day 2, 24 Hours Post-dose | 0.024 (0.012) | 0.022 (0.026)
  Eosinophil; Period 1;Day-1, 24 Hours Pre-dose | 0.136 (0.130) | 0.182 (0.157)
  Eosinophil; Period 1;Day 2, 24 Hours Post-dose | 0.146 (0.130) | 0.204 (0.199)
  Eosinophil; Period 2; Day -1, 24 Hours Pre-dose | 0.231 (0.230) | 0.139 (0.144)
  Eosinophil; Period 2; Day 2, 24 Hours Post-dose | 0.253 (0.245) | 0.156 (0.182)
  Leucocyte; Period 1;Day-1,24 Hours Pre-dose | 5.458 (1.643) | 5.752 (0.907)
  Leucocyte; Period 1;Day 2,24 Hours Post-dose | 5.369 (1.535) | 5.394 (1.019)
  Leucocyte; Period 2;Day -1,24 Hours Pre-dose | 5.736 (1.168) | 5.463 (1.388)
  Leucocyte; Period 2;Day 2,24 Hours Post-dose | 5.887 (1.216) | 5.477 (1.571)
  Lymphocyte; Period 1;Day -1,24 Hours Pre-dose | 2.127 (0.562) | 2.154 (0.493)
  Lymphocyte; Period 1;Day 2,24 Hours Post-dose | 1.916 (0.453) | 2.039 (0.459)
  Lymphocyte; Period 2;Day -1,24 Hours Pre-dose | 2.328 (0.573) | 2.141 (0.409)
  Lymphocyte; Period 2;Day 2,24 Hours Post-dose | 2.186 (0.431) | 1.956 (0.486)
  Monocytes; Period 1;Day -1,24 Hours Pre-dose | 0.480 (0.123) | 0.470 (0.127)
  Monocytes; Period 1;Day 2,24 Hours Post-dose | 0.464 (0.142) | 0.459 (0.125)
  Monocytes; Period 2;Day -1,24 Hours Pre-dose | 0.461 (0.146) | 0.497 (0.126)
  Monocytes; Period 2;Day 2,24 Hours Post-dose | 0.475 (0.160) | 0.457 (0.122)
  Neutrophils;Period 1;Day -1,24 Hours Pre-dose | 2.692 (1.293) | 2.924 (0.706)
  Neutrophils;Period 1;Day 2,24 Hours Post-dose | 2.820 (1.289) | 2.667 (0.667)
  Neutrophils;Period 2;Day -1,24 Hours Pre-dose | 2.691 (0.697) | 2.657 (1.162)
  Neutrophils;Period 2;Day 2,24 Hours Post-dose | 2.949 (0.848) | 2.885 (1.204)
  Platelet; Period 1;Day -1,24 Hours Pre-dose | 288.9 (61.98) | 264.4 (60.63)
  Platelet; Period 1;Day 2,24 Hours Post-dose | 281.2 (65.74) | 244.5 (64.60)
  Platelet; Period 2;Day -1,24 Hours Pre-dose | 264.6 (61.65) | 289.6 (72.29)
  Platelet; Period 2;Day 2,24 Hours Post-dose | 245.0 (56.04) | 274.2 (68.61)

14. Secondary Outcome: Mean Corpuscular Volume (MCV) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of MCV.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Femtoliter
  Period 1; Day -1, 24 Hours Pre-dose | 85.73 (2.834) | 84.86 (4.946)
  Period 1; Day 2, 24 Hours Post-dose | 85.30 (2.796) | 84.50 (4.895)
  Period 2; Day -1, 24 Hours Pre-dose | 84.83 (4.975) | 85.97 (2.903)
  Period 2; Day 2, 24 Hours Post-dose | 84.46 (4.878) | 85.41 (2.847)

15. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of MCH.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Picogram
  Period 1; Day -1, 24 Hours Pre-dose | 29.58 (1.212) | 29.44 (2.140)
  Period 1; Day 2, 24 Hours Post-dose | 29.75 (1.295) | 29.51 (2.190)
  Period 2; Day -1, 24 Hours Pre-dose | 29.40 (2.242) | 29.68 (1.207)
  Period 2; Day 2, 24 Hours Post-dose | 29.54 (2.112) | 29.75 (1.320)

16. Secondary Outcome: Erythrocyte Count at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of erythrocyte count.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
10^12 cells per liter
  Period 1; Day -1, 24 Hours Pre-dose | 5.104 (0.451) | 5.020 (0.480)
  Period 1; Day 2, 24 Hours Post-dose | 4.952 (0.387) | 4.871 (0.424)
  Period 2; Day -1, 24 Hours Pre-dose | 5.006 (0.366) | 4.971 (0.473)
  Period 2; Day 2, 24 Hours Post-dose | 4.838 (0.433) | 4.906 (0.494)

17. Secondary Outcome: Hematocrit at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematocrit.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Proportion of red blood cells in blood
  Period 1; Day -1, 24 Hours Pre-dose | 0.437 (0.036) | 0.426 (0.043)
  Period 1; Day 2, 24 Hours Post-dose | 0.422 (0.033) | 0.411 (0.038)
  Period 2; Day -1, 24 Hours Pre-dose | 0.424 (0.029) | 0.427 (0.040)
  Period 2; Day 2, 24 Hours Post-dose | 0.408 (0.036) | 0.419 (0.041)

18. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Hb) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematology parameters including MCHC and Hb.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Grams per deciliter
  MCHC; Period 1; Day -1, 24 Hours Pre-dose | 34.52 (1.030) | 34.68 (0.957)
  MCHC; Period 1; Day 2, 24 Hours Post-dose | 34.88 (1.084) | 34.89 (1.100)
  MCHC; Period 2; Day -1, 24 Hours Pre-dose | 34.64 (1.100) | 34.54 (0.880)
  MCHC; Period 2; Day 2, 24 Hours Post-dose | 34.95 (1.097) | 34.82 (1.062)
  Hb; Period 1;Day -1, 24 Hours Pre-dose | 15.11 (1.554) | 14.79 (1.833)
  Hb; Period 1;Day 2, 24 Hours Post-dose | 14.74 (1.391) | 14.38 (1.623)
  Hb; Period 2;Day -1, 24 Hours Pre-dose | 14.70 (1.381) | 14.76 (1.591)
  Hb; Period 2;Day 2, 24 Hours Post-dose | 14.29 (1.578) | 14.60 (1.708)

19. Secondary Outcome: Percent Reticulocytes at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of percent reticulocytes.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Percentage of reticulocytes
  Period 1; Day -1, 24 Hours Pre-dose | 1.786 (0.361) | 1.700 (0.346)
  Period 1; Day 2, 24 Hours Post-dose | 1.757 (0.384) | 1.571 (0.297)
  Period 2; Day -1, 24 Hours Pre-dose | 1.729 (0.397) | 1.886 (0.335)
  Period 2; Day 2, 24 Hours Post-dose | 2.350 (2.176) | 1.743 (0.361)

20. Secondary Outcome: Number of Participants With Potential Clinical Importance (PCI) Abnormal Findings for Urinalysis
Description: Urine samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2. PCI ranges for urinalysis parameters were as follows: specific gravity 1.001 to 1.035 kilogram per liter, blood negative (0 to 9) RBC per microliter, pH 4.6 to 8.0, protein negative (0.0 to 0.14) gram per liter, glucose negative (0 to 5.49) millimoles per liter, ketones negative (0.0 to 0.49) millimoles per liter, urobilinogen (0.0 to 1.0) milligrams per deciliter, urine leucocytes negative (0 to 14) leucocytes per microliter, Urine WBC, RBC and epithelial cells 0 to 5 high power per field.
Time Frame: Day -1 and Day 2 of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

21. Secondary Outcome: Respiratory Rate at Indicated Time-points
Description: Respiratory rate of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest.
Time Frame: Day 1 Pre-dose 1.5 hours, Day 1 post-dose 2, 4, and 6 hours and Day 2 post-dose 24 hours of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Breaths per minute
  Period 1; Day 1, 1.5 Hours Pre-dose | 15.0 (1.11) | 15.7 (0.73)
  Period 1; Day 1, 2 Hours Post-dose | 17.3 (2.02) | 17.0 (2.69)
  Period 1; Day 1, 4 Hours Post-dose | 15.5 (2.10) | 14.2 (1.25)
  Period 1; Day 1, 6 Hours Post-dose | 15.0 (2.00) | 14.8 (0.97)
  Period 1; Day 2, 24 Hours Post-dose | 15.9 (2.14) | 16.1 (2.95)
  Period 2; Day 1, 1.5 Hours Pre-dose | 15.8 (1.19) | 15.6 (0.74)
  Period 2; Day 1, 2 Hours Post-dose | 18.4 (1.65) | 18.2 (1.72)
  Period 2; Day 1, 4 Hours Post-dose | 16.7 (3.10) | 18.4 (1.65)
  Period 2; Day 1, 6 Hours Post-dose | 17.9 (1.46) | 19.0 (1.04)
  Period 2; Day 2, 24 Hours Post-dose | 16.2 (1.25) | 16.0 (2.22)

22. Secondary Outcome: Pulse Rate at Indicated Time-points
Description: Pulse rate of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest.
Time Frame: Day 1 Pre-dose 1.5 hours, Day 1 post-dose 2, 4, and 6 hours and Day 2 post-dose 24 hours of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Beats per minute
  Period 1; Day 1, 1.5 Hours Pre-dose | 67.0 (7.95) | 58.1 (8.76)
  Period 1; Day 1, 2 Hours Post-dose | 61.0 (8.17) | 55.1 (8.32)
  Period 1; Day 1, 4 Hours Post-dose | 61.9 (7.44) | 55.6 (7.49)
  Period 1; Day 1, 6 Hours Post-dose | 75.0 (8.74) | 67.2 (12.97)
  Period 1; Day 2, 24 Hours Post-dose | 66.5 (10.26) | 54.3 (7.22)
  Period 2; Day 1, 1.5 Hours Pre-dose | 57.9 (9.08) | 65.1 (6.85)
  Period 2; Day 1, 2 Hours Post-dose | 54.1 (8.88) | 63.1 (8.87)
  Period 2; Day 1, 4 Hours Post-dose | 56.6 (8.67) | 62.8 (7.92)
  Period 2; Day 1, 6 Hours Post-dose | 68.5 (14.09) | 75.1 (8.82)
  Period 2; Day 2, 24 Hours Post-dose | 59.2 (7.59) | 67.1 (8.62)

23. Secondary Outcome: Body Temperature at Indicated Time-points
Description: Body temperature of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest.
Time Frame: Day 1 Pre-dose 1.5 hours, Day 1 post-dose 2, 4, and 6 hours and Day 2 post-dose 24 hours of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Degree Celsius
  Period 1; Day 1, 1.5 Hours Pre-dose | 36.19 (0.305) | 36.27 (0.336)
  Period 1; Day 1, 2 Hours Post-dose | 36.38 (0.333) | 36.23 (0.261)
  Period 1; Day 1, 4 Hours Post-dose | 36.48 (0.336) | 36.59 (0.352)
  Period 1; Day 1, 6 Hours Post-dose | 36.64 (0.303) | 36.79 (0.202)
  Period 1; Day 2, 24 Hours Post-dose | 36.29 (0.317) | 36.24 (0.365)
  Period 2; Day 1, 1.5 Hours Pre-dose | 36.28 (0.372) | 36.29 (0.317)
  Period 2; Day 1, 2 Hours Post-dose | 36.51 (0.400) | 36.42 (0.404)
  Period 2; Day 1, 4 Hours Post-dose | 36.58 (0.347) | 36.51 (0.243)
  Period 2; Day 1, 6 Hours Post-dose | 36.10 (0.421) | 36.63 (0.300)
  Period 2; Day 2, 24 Hours Post-dose | 36.30 (0.321) | 36.11 (0.434)

24. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time-points
Description: Blood pressure of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest.
Time Frame: Day 1 Pre-dose 1.5 hours, Day 1 post-dose 2, 4, and 6 hours and Day 2 post-dose 24 hours of each treatment period
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
Number analyzed (Participants) | 14 | 14
Millimeters of mercury
  SBP, Period 1; Day 1, 1.5 Hours Pre-dose | 110.6 (8.22) | 110.9 (6.39)
  SBP, Period 1; Day 1, 2 Hours Post-dose | 113.4 (7.30) | 111.3 (8.68)
  SBP, Period 1; Day 1, 4 Hours Post-dose | 112.3 (8.39) | 112.1 (4.25)
  SBP, Period 1; Day 1, 6 Hours Post-dose | 111.6 (7.17) | 108.6 (6.46)
  SBP, Period 1; Day 2, 24 Hours Post-dose | 110.9 (6.86) | 115.4 (7.00)
  SBP, Period 2; Day 1, 1.5 Hours Pre-dose | 110.4 (3.97) | 111.2 (10.09)
  SBP, Period 2; Day 1, 2 Hours Post-dose | 113.1 (6.24) | 112.7 (10.94)
  SBP, Period 2; Day 1, 4 Hours Post-dose | 112.6 (8.53) | 111.1 (9.79)
  SBP, Period 2; Day 1, 6 Hours Post-dose | 109.6 (7.14) | 109.5 (8.98)
  SBP, Period 2; Day 2, 24 Hours Post-dose | 113.1 (6.24) | 113.6 (9.05)
  DBP, Period 1; Day 1, 1.5 Hours Pre-dose | 62.9 (6.59) | 64.1 (7.76)
  DBP, Period 1; Day 1, 2 Hours Post-dose | 62.9 (7.69) | 60.9 (6.38)
  DBP, Period 1; Day 1, 4 Hours Post-dose | 62.5 (5.43) | 63.3 (6.94)
  DBP, Period 1; Day 1, 6 Hours Post-dose | 59.3 (3.89) | 59.6 (5.09)
  DBP, Period 1; Day 2, 24 Hours Post-dose | 63.0 (6.80) | 66.2 (7.65)
  DBP, Period 2; Day 1, 1.5 Hours Pre-dose | 111.2 (10.09) | 61.8 (7.20)
  DBP, Period 2; Day 1, 2 Hours Post-dose | 66.2 (7.65) | 63.1 (9.12)
  DBP, Period 2; Day 1, 4 Hours Post-dose | 63.5 (8.55) | 62.6 (8.21)
  DBP, Period 2; Day 1, 6 Hours Post-dose | 59.4 (4.97) | 60.2 (7.79)
  DBP, Period 2; Day 2, 24 Hours Post-dose | 63.9 (7.41) | 67.7 (7.90)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and Non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to Day 16 in each treatment period.
Description: SAEs and Non-SAEs were reported by treatment for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment.
Arm/Group | SKF101804 Cefixime | Cefixime Reference Formulation
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT03408392/Prot_SAP_000.pdf